CLINICAL TRIAL: NCT06391736
Title: A Multi-centered, Single Arm, Open Labeled, Study to Evaluate the Safety, Tolerability, and Efficacy of an Adeno-associated Virus Vector Expressing the Human Acid Alpha-glucosidase (GAA) Transgene Intravenous Injection in Patients With Late-onset Pompe Disease
Brief Title: Evaluation of the Safety and Efficacy of Late-onset Pompe Disease Gene Therapy Drug
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GeneCradle Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JLJY-GC301-LOPD-001
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Pompe Disease (Late-onset)
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dosage group (Experimental): Single intravenous administration of GC301 at a dose of 3.0 x 10^13 vector genomes per kilogram body weight
  Interventions: Genetic: GC301
- High dosage group (Experimental): Single intravenous administration of GC301 at a dose of 6.0 x 10^13 vector genomes per kilogram body weight
  Interventions: Genetic: GC301

INTERVENTIONS:
Genetic: GC301 — GC301, is an adeno-associated virus 9 (AAV9) vector delivering a functional copy of the human GAA gene

SUMMARY:
This study is being conducted to evaluate the safety and effectiveness of GC301 adeno-associated virus vector expressing codon-optimized human acid alpha-glucosidase (GAA) as potential gene therapy for Pompe disease. Patients diagnosed with late-onset Pompe disease （LOPD） who are ≥ 6 years old will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 years, males or females;
* Patient has a diagnosis of LOPD;
* Patient has upright FVC ≥ 30% of predicted normal value;
* A 6MWT ≥ 40 meters, assistive device allowed;
* The patient's legal guardian(s) must be able to understand the purpose and risks of the study and voluntarily provide signed and dated informed consent prior to any study-related procedures being performed.

Exclusion Criteria:

* Patient who has any history or concurrent clinical organic disease, including cardiovascular and liver diseases, respiratory system, nervous system disease, or any other condition that, in the opinion of the investigator, makes the subject unsuitable for participation in the study.
* Patient who requires invasive mechanical ventilation, or rely on noninvasive non-non-invasive assisted ventilation when sitting upright;
* Patient who is positive for human immunodeficiency (HIV) antibody, hepatitis B surface antigen, hepatitis C antibody, or treponema pallidum antibody;
* Patient with a history of glucocorticoid allergy;
* Patient who has a contraindication to study drug or to corticosteroids, or has demonstrated hypersensitivity to any of the components of the study drug;
* Patient who has AAV9 neutralizing antibody titer ≥ 1:100；
* Patient who has participated in a previous gene therapy research trial;
* Pregnant or lactating female participants;
* Patients who have fertility plans within 6 months from screening to the end of the study and are unwilling to take effective physical contraceptive measures (such as a condom, intrauterine device, contraceptive ring, ligation, abstinence, etc.) for contraception (including the subject's partner);

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | 52 weeks
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability
Dose-limiting toxicity (DLT) rate based on protocol-specific adverse events (Phase 1) | within 30 days after treatment
Percent Predicted Upright Forced Vital Capacity (FVC)(Phase 2) | 52 weeks
  Change from baseline in percentage of predicted FVC measured by pulmonary function testing

SECONDARY OUTCOMES:
6-Minute Walk Test | 52 weeks
  Change from baseline in the distance walked in the 6 minute walk test (6MWT), which is a standardized assessment of how far an individual can walk on a hard, flat surface in a period of 6 minutes
Maximum Inspiratory Pressure (MIP) | 52 weeks
  Change from baseline in MIP measured by pulmonary function testing
Maximum Expiratory Pressure (MEP) | 52 weeks
  Change from baseline in MEP measured by pulmonary function testing
Muscle Status Testing - Quick Motor Function Test (QMFT) Measure | 52 weeks
  Measurement of functional motor abilities using the Quick Motor Function Test (QMFT) will be performed and the results compared with baseline.
Quality of life evaluation: 12-item short form health survey (SF-12) for LOPD participants | 52 weeks
  SF-12, a 12 item-questionnaire, used to assess health-related quality of life in participants aged >=18 years at screening/baseline. SF-12 consisted of 12 items, which were categorized into eight domains (subscales) of functioning and well-being: physical functioning, role-physical, role emotional, mental health, bodily pain, general health, vitality and social functioning, with each domain score ranged from 0 (poor health) to 100 (better health), higher scores indicated good health condition. These eight domains were further summarized into 2 summary scores, physical component summary (PCS) and mental component summary (MCS). The score range for each of these 2 summary scores was from 0 (poor health) to 100 (better health), higher scores indicated a better health-related quality of life.
Time needed for non-invasive ventilatory support | 52 weeks
  Change from baseline in time duration that needed for non-invasive ventilatory support
The viral load of adeno-associated virus (AAV) vector | 52 weeks
  To assess the change of AAV vector copy numbers within 52 weeks after administration.
Occurrence of immune response against AAV capsid annd GAA transgene | 52 weeks

OTHER OUTCOMES:
GAA enzymatic activity | 52 weeks
  Change from baseline in GAA enzymatic activity in muscle biopsies
GAA enzymatic activity | 52 weeks
  Change from baseline in GAA enzymatic activity in blood
Glycogen content in muscle | 52 weeks
  Change from baseline in glycogen content in muscle biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Guang Yang, Study Chair — Chinese PLA General Hospital; Guang Yang, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China